CLINICAL TRIAL: NCT02157324
Title: A Multicenter, Open-label, Phase 1 Pilot Study of ACP-196 in Combination With ACP-319 in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: Acalabrutinib in Combination With ACP-319, for Treatment of Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-CL-002
Record Dates: First submitted 2014-05-30; First posted 2014-06-06 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Bruton tyrosine kinase inhibitor; Btk
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; N-(1-(7-fluoro-2-(pyridin-2-yl)quinolin-3-yl)ethyl)-9H-purin-6-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acalabrutinib (Experimental): Starts with acalabrutinib for 7 days, then combined with ACP-319 afterwards.
  Interventions: Drug: acalabrutinib; Drug: ACP-319
- ACP-319 (Experimental): Starts with ACP-319 for 7 days, then combined with acalabrutinib afterwards.
  Interventions: Drug: acalabrutinib; Drug: ACP-319

INTERVENTIONS:
Drug: acalabrutinib
  Other Names: ACP-196
Drug: ACP-319

SUMMARY:
This study is evaluating the safety and efficacy of the combined use of acalabrutinib and ACP-319, for the treatment of chronic lymphocytic leukemia (CLL)

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age with a confirmed diagnosis of CLL, which has relapsed after, or been refractory to, ≥ 1 previous treatments for CLL; however, subjects with 17p deletion are eligible if they have relapsed after, or been refractory to, 1 prior treatment for CLL.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use contraception during the study and for 30 days after the last dose of study drugs if sexually active and able to bear or beget children.

Exclusion Criteria:

* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years.
* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib and/or ACP-319, or put the study outcomes at undue risk.
* Significant cardiovascular disease.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Any immunotherapy within 4 weeks of first dose of study drug.
* For subjects with recent chemotherapy or experimental therapy the first dose of study drug must occur after 5 times the half-life of the agent(s).
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation.
* Ongoing immunosuppressive therapy, including systemic or enteric corticosteroids for treatment of CLL or other conditions. Note: Subjects may be using topical or inhaled corticosteroids as therapy for comorbid conditions.
* Central nervous system (CNS) involvement by CLL.
* Grade ≥ 2 toxicity (other than alopecia).
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) or any uncontrolled active systemic infection.
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
* Absolute neutrophil count (ANC) < 0.75 x 109/L or platelet count < 50 x 109/L unless due to disease involvement in the bone marrow.
* Creatinine > 1.5 x institutional upper limit of normal (ULN); total bilirubin > 1.5 x ULN (unless due to Gilbert's disease); and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN unless disease related.
* Significant screening ECG abnormalities including left bundle branch block, 2nd degree AV block type II, 3rd degree block, Grade 2 or higher bradycardia, and QTc > 480 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date of randomization until the day of documented progression or date of death from any cause, whichever came first, assessed up to 60 cycles of 28 days.
  The frequency (number and percentage) of treatment-emergent AEs will be reported in each treatment group by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class and Preferred Term. Summaries will also be presented by the severity of the AE (per CTCAE, v4.03) and by relationship to study drug.

SECONDARY OUTCOMES:
Drug Exposure, Area Under the Plasma Concentration-time Curve | From 30 min before first dose to day-28 of cycle-6 of a 28 day cycle
  PK sample schedule: Cycle 1 - Up to 30 minutes before dosing and 0.5, 1, 2, 4, 6, 12, 13, and 24 hours after the morning dose of Day 1 and 28. Also, 30 min before morning dose of cycle 1 - day 8,15 & 22, cycle 2 - day 15 & 28, and cycle 3 to 6 - day 28.
Drug Exposure, Maximum observed plasma concentration | From 30 min before first dose to 30 min before day-28 of cycle-6 of 28 day cycles
  PK sample schedule: Cycle 1 - Up to 30 minutes before dosing and 0.5, 1, 2, 4, 6, 12, 13, and 24 hours after the morning dose of Day 1 and 28. Also, 30 min before morning dose of cycle 1 - day 8,15 & 22, cycle 2 - day 15 & 28, and cycle 3 to 6 - day 28.
Drug Exposure, Time of the maximum plasma concentration | From 30 min before first dose till 30 before day-28 of cycle-6 of 28 day cycles
  PK sample schedule: Cycle 1 - Up to 30 minutes before dosing and 0.5, 1, 2, 4, 6, 12, 13, and 24 hours after the morning dose of Day 1 and 28. Also, 30 min before morning dose of cycle 1 - day 8,15 & 22, cycle 2 - day 15 & 28, and cycle 3 to 6 - day 28.
Overall Response rate | Pretreatment, then end of cycles 2, 4, 9, 12, 18 and then every 6 cycles to cycle 36. After that at cycle 48 and 60 of 28 day cycles.
  A CT scan with contrast (unless contraindicated) of the neck, chest, abdomen, and pelvis and any other disease sites are required for the pretreatment tumor assessment.
Duration of Response | Pretreatment, then end of cycles 2, 4, 9, 12, 18 and then every 6 cycles to cycle 36. After that at cycle 48 and 60 of 28 day cycles.
  The duration of response is measured from the time measurement criteria are met for Complete Response or Partial Response (whichever is first recorded) until the first date that recurrent disease or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the study treatment started). Kaplan-Meier methodology will be used to estimate event-free curves and corresponding quantiles (including the median).
Progression-Free Survival | Pretreatment, then end of cycles 2, 4, 9, 12, 18 and then every 6 cycles to cycle 36. After that at cycle 48 and 60 of 28 day cycles.
  PFS is measured from the time of first study drug administration until the first date that recurrent disease or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the study treatment started). Kaplan-Meier methodology will be used to estimate the event-free curves and corresponding quantiles (including the median).

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613 acertamc@dlss.com
Locations (3):
- United States (3):
  - Research Site, Columbus, Ohio
  - Research Site, Hermitage, Tennessee
  - Research Site, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home